CLINICAL TRIAL: NCT03689556
Title: A Phase II Clinical Trial Evaluating the Role of FLT PET/CT in Predicting Treatment Response of Carbon-ion Radiotherapy for Patients With Locoregionally Recurrent Nasopharyngeal Carcinoma
Brief Title: Examine the Prognostic Role of FLT PET/CT for Patients With LR-NPC Treated by Carbon Ion Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Jiade J. Lu, Professor, Shanghai Proton and Heavy Ion Center
Other Study IDs: SPHIC-TR-HNCNS-2018-19
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Recurrent Nasopharyngeal Carcinoma
Keywords: FLT PET/CT; carbon ion radiation therapy; re-irradiation
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FLT PET/CT: Patients with locoregionally recurrent nasopharyngeal carcinoma (LR-NPC) will receive FLT PET/CT scans before CIRT and after completion of CIRT.
  Interventions: Diagnostic Test: FLT PET/CT

INTERVENTIONS:
Diagnostic Test: FLT PET/CT — Patients will receive 3'-deoxy-3'-[18F]fluorothymidine (FLT) PET/CT scans before CIRT and after completion of CIRT.

SUMMARY:
We aim, in this study, to examine whether reduction of FLT PET derived SUV before and after carbon ion radiotherapy can predict the treatment response and survivals for patients with locoregionally recurrent nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
This is a single-arm phase II clinical trial evaluating the prognostic value of FLT PET/CT for patients with locoregionally recurrent nasopharyngeal carcinoma. All patients will receive FLT PET/CT scans before and after carbon ion radiotherapy (CIRT). The sensitivity and specificity of reduction of FLT uptake reduction in terms of predicting the treatment outcome evaluated by MRI at 3 months after completion of CIRT according to RECIST 1.1. Its predictive value of OS, LPFS, RPFS and DMFS will be examined as well.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed as primary nasopharyngeal carcinoma;
* With recurrence at nasopharynx and/or recurrent retropharyngeal lymph node, recurrence was diagnosed by imaging or pathology studies;
* Already received one course of definitive radiation therapy, at least 6 months ago;
* Able to receive contrast MRI scan and PET/CT scan;
* ECOG: 0-2;
* Anticipated survival time >= 12 months;
* With sufficient major organ functions;
* Willing to sign informed consent.

Exclusion Criteria:

* Metal implants that might significantly influence the radiation dose distribution;
* Dose constrains for organs-at-risk are beyond acceptable limit;
* With comorbidities/conditions that might influence the effectiveness of carbon-ion therapy;
* Pregnant or within lactation period;
* Drug/alcohol addiction;
* With mental disorder that might impede the completion of therapy.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive LR-NPC patients treated at SPHIC will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity | The reduction of FLT uptake will be calculated over two time points, at the baseline and at the time point that CIRT is completed.
  The sensitivity and specificity of FLT uptake reduction in predicting the treatment response evaluated by MRI scan at 3 months after completion of CIRT.

SECONDARY OUTCOMES:
Overall survival (OS) | Duration from the date the diagnosis of LR-NPC is made until date of patient death or the last follow-up, whichever comes first, assessed up to 36 months
  3-year overall survival
Local progression-free survival (LPFS) | Duration from the date the diagnosis of LR-NPC is made until date of documented local failure or the last follow-up/patient death, whichever comes first, assessed up to 36 months
  3-year local progression-free survival
Regional progression-free survival (RPFS) | Duration from the date the diagnosis of LR-NPC is made until date of documented regional failure or the last follow-up/patient death, whichever comes first, assessed up to 36 months
  3-year regional progression-free survival
Distant metastasis-free survival (DMFS) | Duration from the date the diagnosis of LR-NPC is made until date of documented distant metastasis or the last follow-up/patient death, whichever comes first, assessed up to 36 months
  3-year distant metastasis-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Jiade J Lu, MD, Principal Investigator — Shanghai Proton and Heavy Ion Center,Shanghai, SPHIC

IPD SHARING:
Plan to Share IPD: Undecided